CLINICAL TRIAL: NCT01578902
Title: Hypofractionated Accelerated Radiotherapy for Low Risk Localized Prostate Cancer (pHART 3)
Brief Title: Hypofractionated Accelerated Radiotherapy for Low Risk Localized Prostate Cancer
Acronym: pHART3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Association of Radiation Oncology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 371-2006
Record Dates: First submitted 2011-10-31; First posted 2012-04-17 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Prostate Cancer
Keywords: Prostatic Neoplasms; Radiotherapy; Hypofractionation; Low Risk Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hypofractionated radiotherapy using SABR (Experimental): Stereotactic radiation: 35Gy in 5 fractions over 29 days
  Interventions: Radiation: Stereotactic ablative body radiotherapy

INTERVENTIONS:
Radiation: Stereotactic ablative body radiotherapy — 35Gy/5 fractions/29 days
  Other Names: standard linear accelerator delivery

SUMMARY:
The purpose of this study is to determine the safety and efficacy of a short course of radiotherapy (35 Gy / 5 fractions / 29 days) for the treatment of low-risk prostate cancer.

DETAILED DESCRIPTION:
Rationale for Proposed Study With the availability of intensity modulated radiotherapy (IMRT) at the Odette Cancer Centre (OCC), there is an opportunity to explore the use of a much more intensive hypofractionation schedule for prostate cancer. Using an alpha/beta ratio of 1.3, a dose of 35 Gy in 5 fractions would be equivalent to 88 Gy delivered in 2 Gy fractions. For normal tissues (alpha/beta value of 2), this would be equivalent to 78 Gy in 2 Gy fractions. As such, the linear quadratic equation predicts that 35 Gy in 5 fractions should not result in any increased late toxicity for normal tissues compared to standard dose escalated radiotherapy. However, the biological dose to the prostate cancer would be significantly increased. As a safety precaution for this study proposal, the investigators propose to deliver 35 Gy in 5 fractions over 5 weeks (one radiotherapy fraction of 7 Gy per week) to allow for normal tissue repair.

With IMRT, it is expected that there will be superior conformality of the high dose region around the target volume. As well, the use of daily on-line imaging will allow us to eliminate interfraction prostate motion errors and use tighter planning target volume margins for any residual intrafraction motion. At OCC, such an approach has already been shown to be feasible and is currently employed in the phase 1/2 concomitant boost study for high risk prostate cancer.

If proven to be safe and effective, such a hypofractionated radiotherapy schedule may have significant practical advantages as well. With only 1 fraction of radiotherapy delivered each week (for a total of 5 weeks), there are huge savings in resource utilization and increased convenience for patients.

The investigators propose to start a small phase 1 study to explore the use of this dose fractionation for men with low risk prostate cancer. The primary endpoint for this small pilot study would be acute and late normal tissue toxicities. If proven to be feasible and safe, external peer-reviewed funding will be sought to further explore this novel treatment schedule in a larger phase 2 setting.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed (Appendix A)
* Adult men greater than 18 years of age
* Histologically confirmed diagnosis of adenocarcinoma of the prostate (centrally reviewed).
* Clinical stage T1-T2b, Gleason Score < 6, and PSA < 10 ng/mL
* Less than 50% of biopsy cores +ve for cancer
* Less than 50% overall surface area involved with cancer
* Neoadjuvant hormone suppression therapy is allowed. However, PSA, must have been performed within 2 months of starting androgen suppression therapy. If androgen suppression therapy has been started LHRH agonist must be continued for a minimum of 3 months before initiation of gold fiducial marker insertion & radiotherapy planning.

Exclusion Criteria:

* Prior pelvic radiotherapy.
* Concurrent anticoagulation medication (if it is unsafe to discontinue for gold seed insertion)
* Diagnosis of bleeding diathesis
* Presence of a hip prosthesis
* Pelvic girth >40cm (to ensure visibility of gold seeds on electronic portal imaging device)
* Large prostate (> 60 cm3) on imaging
* Severe lower urinary tract symptoms (International Prostate Symptom Score > 15 or nocturia > 3)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2006-10; Primary Completion 2008-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Loblaw, MD, Principal Investigator — Sunnybrook Health Sciences Centre; Patrick Cheung, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Quon HC, Musunuru HB, Cheung P, Pang G, Mamedov A, D'Alimonte L, Deabreu A, Zhang L, Loblaw A. Dose-Escalated Stereotactic Body Radiation Therapy for Prostate Cancer: Quality-of-Life Comparison of Two Prospective Trials. Front Oncol. 2016 Aug 29;6:185. doi: 10.3389/fonc.2016.00185. eCollection 2016. PMID 27622157

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were prospectively recruited from the Odette Cancer Centre from Oct 2006 to July 2008.
Groups:
- Hypofractionated Radiation: 35 Gy in 5 fractions of image-guided intensity modulated radiotherapy (IGRT) delivered over 29 days.
  Hypofractionated radiotherapy: 35Gy/5 fractions/29 days
Period: Overall Study
Arm/Group | Hypofractionated Radiation
Started | 84
Completed | 84
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Patients: Inclusion criteria were men over 18 years of age with histologically confirmed diagnosis of adenocarcinoma of the prostate. Only patients with clinical stage T1-T2b (TNM 2002) [18] Gleason Sum 66 and PSA 610 ng/ml were eligible. Neoadjuvant androgen deprivation therapy (ADT) was allowed for cytoreduction. Patients were excluded if they had prior pelvic radiation therapy, a bleeding diathesis which precluded safe gold seed insertion, the presence of hip prosthesis or pelvic girth >40 cm. Lastly, prostate size >90cm3 on imaging or severe lower urinary tract symptoms (IPSS > 19)
Arm/Group | All Patients
Number analyzed (Participants) | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 44
Age, Continuous [Median (Full Range); unit: years] | 67 [42 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 84
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 84

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Grade 3+ Gastrointestinal Toxicity
Description: Common Terminology Criteria for Adverse Events (CTCAE) v3.0
Time Frame: Acute period (up to 6 months)
Measure: Number; unit: participants
Groups:
- Hypofractionated Radiation: 35 Gy in 5 fractions of image-guided intensity modulated radiotherapy (IGRT) delivered over 29 days.
  The co-primary outcome variable (Grade 3+ acute gastrointestinal toxicity) was observed in 0% of patients.
Arm/Group | Hypofractionated Radiation
Number analyzed (Participants) | 84
participants | 0

2. Secondary Outcome: Incidence of Grade 3+ Genitourinary Toxicity
Description: Common Terminology Criteria for Adverse Events (CTCAE) v3.0
Time Frame: Acute (up to 6 months) and Late (6 months and after)
Measure: Count of Participants; unit: Participants
Groups:
- Hypofractionated Radiation: 35 Gy in 5 fractions of image-guided intensity modulated radiotherapy (IGRT) delivered over 29 days.
  The co-primary endpoint (Grade 3+ acute genitourinary toxicity) was observed in 1% (1/84) patients.
Arm/Group | Hypofractionated Radiation
Number analyzed (Participants) | 84
Participants | 1

3. Secondary Outcome: Incidence of Grade 3+ Rectal and Urinary Toxicity
Description: Common Terminology Criteria for Adverse Events (CTCAE) v3.0
Time Frame: Late (6 months and after)
Population: low risk prostate cancer patients were treated with SABR 35Gy in 5 fractions over 29 days
Measure: Number; unit: participants
Arm/Group | Hypofractionated Radiation
Number analyzed (Participants) | 84
participants
  Acute GU grade 3+ toxicity | 1
  Acute GI grade 3+ toxicity | 0
  Late GU grade 3+ toxicity | 0
  Late GI grade 3+ toxicity | 1

4. Secondary Outcome: Patient Reported Quality of Life
Description: Expanded Prostate Cancer Index Composite (EPIC)
Time Frame: up to 5 years
Population: Patients were low risk prostate cancer patients treated with SABR 35Gy in 5 fractions over 29 days.
Measure: Number; unit: percentage with change in QOL
Arm/Group | Hypofractionated Radiotherapy Using SABR
Number analyzed (Participants) | 84
percentage with change in QOL
  Bowel quality of life change | 22
  Bladder quality of life change | 16
  Sexual quality of life change | 33

5. Secondary Outcome: Biochemical (ie. Prostate Specific Antigen) Disease Free Survival
Description: Failure = Follow-up PSA greater than nadir PSA + 2 ng/ml
Time Frame: 5 year
Population: low risk prostate cancer patients treated with SABR 35 Gy in 5 fractions over 29 days
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Hypofractionated Radiation
Number analyzed (Participants) | 84
percent | 96 [91.5 to 100]

6. Secondary Outcome: Biopsy Positive Rate
Description: Patients were biopsied at 3 years post treatment
Time Frame: 3 year
Population: low risk prostate cancer patients treated with SABR 35 Gy in 5 fractions over 29 days
Measure: Count of Participants; unit: Participants
Arm/Group | Hypofractionated Radiation
Number analyzed (Participants) | 84
Participants | 3

ADVERSE EVENTS:
Arm/Group | Hypofractionated Radiation
Serious Adverse Events (participants affected / at risk) | 2/84
Other Adverse Events (participants affected / at risk) | 34/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypofractionated Radiation (N=84)
acute urinary retention (Renal and urinary disorders) | 1 (1)
rectalcutaneous fistula (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypofractionated Radiation (N=84)
acute grade 2 genitourinary (Renal and urinary disorders) | 16 (16)
acute grade 2 gastrointestinal toxicity (Gastrointestinal disorders) | 8 (8)
late grade 2 gastrointestinal toxicity (Gastrointestinal disorders) | 6 (6)
late grade 2 genitourinary toxicity (Renal and urinary disorders) | 5 (5)
late grade 3+ GI toxicity (Gastrointestinal disorders) | 1 (1)
late grade 3+ GU toxicity (Renal and urinary disorders) | 0 (0)
acute grade 3+ GU toxicity (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No